CLINICAL TRIAL: NCT04309747
Title: A Prospective, Multicenter Clinical Trial of Safety and Effectiveness of Nanosecond Knife Ablation for Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Tian'an Jiang, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nanosecond001; nanosecond knife01 (Registry Identifier: nanosecond knife tumor ablation for liver cancer)
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Liver Cancer
Keywords: nanosecond knife; liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: To evaluate whether the nanosecond knife can achieve the effectiveness and safety of liver cancer ablation treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nanosecond knife group (Experimental): This trial is a prospective, multi-center, single-arm clinical trial. Four hospitals with national medical clinical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive nanosecond pulse ablation therapy according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the product will be made according to groups.
  Interventions: Procedure: nanosecond knife liver cancer ablation

INTERVENTIONS:
Procedure: nanosecond knife liver cancer ablation — This trial is a prospective, multi-center, single-arm clinical trial. Four hospitals with national medical clinical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive nanosecond pulse ablation therapy according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the product will be made according to groups.

SUMMARY:
This is a prospective, multi-center, single-arm clinical trial. Four hospitals with national medical clinical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive nanosecond pulse ablation therapy according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the product will be made according to groups.

DETAILED DESCRIPTION:
The prospective, multi-center, single-arm clinical trial is to evaluate whether the nanosecond knife can achieve the effectiveness and safety of liver cancer ablation treatment. Four hospitals with national medical clinical trial institution qualifications are selected as clinical trial centers. This clinical trial requires 190 subjects. Qualified participants will receive nanosecond pulse ablation therapy according to the routine procedures. The results will be recorded according to the requirements of the primary outcome (the effective rate of nanosecond knife ablation for liver cancer) and secondary outcomes (partial response rate, secondary ablation rate, progression-free survival, overall survival rate, quality of life score, alpha-fetoprotein levels, technical success rate, local control rate, complication rate, device Use satisfaction of nanosecond knife ablation for liver cancer). The first 2-month follow-up after the operation, CT, MR, CEUS, liver function, tumor markers were reviewed monthly to observe the lesion necrosis and tumor marker changes. After that, tumor markers, CEUS, or three-phase CT/MRI of liver were examined every 2 to 3 months. After two years, tumor markers, CEUS, or three-phase CT/MRI of liver were examined every 3 to 6 months. After then, statistical comparisons of effectiveness and safety of the product will be made according to groups.

ELIGIBILITY:
Inclusion Criteria:

1. Liver malignant tumors with clear histopathology and cytology, or liver malignant tumors that meet clinical diagnosis and staging criteria.
2. Age: 18-75 years old, regardless of gender.
3. Liver function: Child-Pugh A or B, or Child C will reach B.
4. No serious heart, lung, brain and other organ dysfunction. Normal or nearly normal blood coagulation function. Prothrombin time does not exceed 50% of the normal control, and platelets are more than 50 × 109 / L.
5. It is usually suitable for single tumor with a maximum diameter of ≤5cm, or the number of tumors of ≤3 and a maximum diameter of ≤3cm.
6. For single tumors > 5 cm in diameter that cannot be surgically removed, or multiple tumors with a maximum diameter > 3 cm, local ablation can be used as p palliative comprehensive treatment.
7. According to CT and MRI, there are no macrovascular and bile duct invasions visible by the naked eye.
8. Patients signed informed consent to participate in the trial.

Exclusion Criteria:

1. The lesion of liver cancer is huge or diffuse ;
2. Merged portal vein to secondary branch tumor thrombus or hepatic vein tumor thrombus, invasion of nearby organs or distant metastasis;
3. tumors located on the surface of the liver, of which more than 1/3 tumor size are bare;
4. liver function: Child-pugh C, those could not improve after liver protective treatment;
5. Esophageal (bottom of stomach) varices rupture and bleeding within 1 month before treatment;
6. Uncorrectable coagulation dysfunction and severe haematological abnormalities, who tend to severe bleeding;
7. Refractory large amount of ascites and cachexia;
8. active infection, especially inflammation of the biliary system;
9. Severe failure of major organs such as liver, kidney, heart, lung and brain;
10. Patients with unconsciousness or unable to cooperate with treatment;
11. Subjects could not be followed up and fell off;
12. Those who discontinued treatment, or the case records were incomplete for various reasons, and were determined by researchers to be unable to be evaluated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness analysis | 12 months
  The effective rate of nanosecond knife ablation for liver cancer

SECONDARY OUTCOMES:
Secondary validity analysis | 12 months
  partial response rate of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  secondary ablation rate of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  progression-free survival of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  overall survival rate of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  quality of life score of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  alpha-fetoprotein levels
Secondary validity analysis | 12 months
  technical success rate of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  local control rate of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  complication rate of nanosecond knife ablation for liver cancer
Secondary validity analysis | 12 months
  device Use satisfaction of nanosecond knife ablation for liver cancer

IPD SHARING:
Plan to Share IPD: Yes
This trial is a prospective, multi-center, single-arm clinical trial. Four hospitals with national medical clinical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive nanosecond pulse ablation therapy according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the product will be made according to groups.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Gu YK, Luo RG, Huang JH, Si Tu QJ, Li XX, Gao F. Transarterial embolization ablation of hepatocellular carcinoma with a lipiodol-ethanol mixture. World J Gastroenterol. 2010 Dec 7;16(45):5766-72. doi: 10.3748/wjg.v16.i45.5766. PMID 21128329
- [Background] Bargellini I, Vignali C, Cioni R, Petruzzi P, Cicorelli A, Campani D, De Simone P, Filipponi F, Bartolozzi C. Hepatocellular carcinoma: CT for tumor response after transarterial chemoembolization in patients exceeding Milan criteria--selection parameter for liver transplantation. Radiology. 2010 Apr;255(1):289-300. doi: 10.1148/radiol.09090927. PMID 20308465
- [Background] Fruhling P, Nilsson A, Duraj F, Haglund U, Noren A. Single-center nonrandomized clinical trial to assess the safety and efficacy of irreversible electroporation (IRE) ablation of liver tumors in humans: Short to mid-term results. Eur J Surg Oncol. 2017 Apr;43(4):751-757. doi: 10.1016/j.ejso.2016.12.004. Epub 2017 Jan 11. PMID 28109674
- [Background] Distelmaier M, Barabasch A, Heil P, Kraemer NA, Isfort P, Keil S, Kuhl CK, Bruners P. Midterm Safety and Efficacy of Irreversible Electroporation of Malignant Liver Tumors Located Close to Major Portal or Hepatic Veins. Radiology. 2017 Dec;285(3):1023-1031. doi: 10.1148/radiol.2017161561. Epub 2017 Aug 11. PMID 28799842
- [Background] Bruix J, Sherman M, Llovet JM, Beaugrand M, Lencioni R, Burroughs AK, Christensen E, Pagliaro L, Colombo M, Rodes J; EASL Panel of Experts on HCC. Clinical management of hepatocellular carcinoma. Conclusions of the Barcelona-2000 EASL conference. European Association for the Study of the Liver. J Hepatol. 2001 Sep;35(3):421-30. doi: 10.1016/s0168-8278(01)00130-1. No abstract available. PMID 11592607
- [Derived] Liu J, Fang C, Jin X, Tian G, Sun Z, Hong L, Pan J, Chen X, Zhao J, Cao H, Jiang T. Nanosecond pulsed electric field ablation-induced modulation of sphingolipid metabolism is associated with Ly6c2+ mononuclear phagocyte differentiation in liver cancer. Mol Oncol. 2023 Jun;17(6):1093-1111. doi: 10.1002/1878-0261.13372. Epub 2023 Jan 21. PMID 36587393
- [Derived] Xu M, Xu D, Dong G, Ren Z, Zhang W, Aji T, Zhao Q, Chen X, Jiang T. The Safety and Efficacy of Nanosecond Pulsed Electric Field in Patients With Hepatocellular Carcinoma: A Prospective Phase 1 Clinical Study Protocol. Front Oncol. 2022 Jul 13;12:869316. doi: 10.3389/fonc.2022.869316. eCollection 2022. PMID 35912221